CLINICAL TRIAL: NCT07227701
Title: A Comparison of Satiety Effects of High Protein Snack Bars and High Carbohydrate Snack Bars
Brief Title: A Comparison of Satiety Effects Two Commercially Available Snack Bars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Bret McConaughy Rust, Principal Investigator, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Snacks and Satiety; Linus Technology (Other: Linus Technology)
Record Dates: First submitted 2025-08-25; First posted 2025-11-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Satiety
Keywords: Satiety; Hunger; food intake; satisfaction; desire to eat; snack bars
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Acute, single blinded, randomized crossover design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two high carbohydrate snack bars conferring 150 Kcal each for a total of 300 Kcal. (Active Comparator): The snack bars are presented with ad libitum bottled water.
  Interventions: Other: High carbohydrate snack bar
- Two high protein snack bars conferring 150 Kcal each for a total of 300 Kcal. (Experimental): This arm involves a snack bar with a different nutrient profile than the comparator.
  Interventions: Other: High protein snack bar

INTERVENTIONS:
Other: High carbohydrate snack bar — A snack bar containing 26 grams of carbohydrate and 2 grams of protein.
  Arms: Two high carbohydrate snack bars conferring 150 Kcal each for a total of 300 Kcal.
Other: High protein snack bar — A snack bar containing 28 grams of protein and 2 grams of carbohydrate
  Arms: Two high protein snack bars conferring 150 Kcal each for a total of 300 Kcal.

SUMMARY:
The researchers are investigating the satiety effects of two commercially available snack bars. Qualified participants are age 18-65 with a body mass index of 18.5 to 29.9 kilograms of body weight per meter squared in height who are in good metabolic health. Participants will engage in two study visits conducted at the Indiana University--Bloomington Innovation Center.

Study visits are separated by a 1-14 day washout period. Prior to each study visit, participants are asked to engage in normal activity and to refrain from strenuous exercise. Furthermore, subjects are asked to consume a typical diet the day prior to the study visit with one caveat; they are to consume standard frozen dinners (evening meal) of their choosing between 7-8 PM and to remain fasted afterward except for water and non-caloric beverages until the study visit the following day. The amount of food provided for the evening meal is estimated using a standard calorie calculator based on the Mifflin-St. Jeor equation and an estimate of their activity level. Subjects are instructed to consume only as much of the provided food as needed to become comfortably full as they would ordinarily. Subjects record their diet for the day.

Upon arrival at the Innovation Center between 8-8:40 AM, compliance with the prior day protocol is verified through interview, and the diet record is reviewed. Participants consume 300 kcal of snack bars and complete visual analogue scales to assess hunger, fullness, desire to eat, and satisfaction at fasting and at 30 minute intervals from the fasting measurement for 2 hours. Immediately after consuming the snack bars, subjects complete a sensory evaluation of the snack bars. Fifteen to thirty minutes after completion of the final visual analogue scale, subjects will be presented with an individual buffet which they consume ad libitum until comfortably full.

A second study visit that mirrors the first but with different bars is conducted after the washout period (1-14 days).

DETAILED DESCRIPTION:
The study protocol is initiated after enrollment with a Food Frequency Questionnaire and a Three-factor eating questionnaire conducted during the screening visit after the participant's qualifications have been verified. After the questionnaires have been completed, the study visits and food pick ups are scheduled according to the availability of the subject and the study calendar. At the end of the screening appointment, the subject selects the frozen dinners to be consumed the evening prior to the study visit.

The study is a crossover design in which investigators will assess the immediate effects of a single meal of two commercially available snack bars on subjective feelings of satiety over 2 hours and on energy and nutrient intake from a subsequent meal 2:15 to 2:30 following consumption of the bars. Study visits will be scheduled between 1 and 14 days apart.

Subjects will consume a standard meal between 7 and 8 PM the evening prior to each study visit and complete a satiety questionnaire after finishing the meal. The subjects record all food consumed the day prior to the study visit including the dinner meals provided by the study. Participants will pick up food at the Indiana University-Bloomington School of Public Health the day prior to the scheduled study visits. This visit consists of dispensing the evening meals in lunch coolers packed with icepacks and the frozen meals the participant selected in the screening appointment. The study visit protocol for the following day is reviewed briefly. Appointment reminders are set up as emails and calendar invitations instructing the participant to consume the meals between 7-8 PM that night, to complete a satiety questionnaire, the link to which is embedded in the emails, and to remain fasted except for water and non-caloric beverages until the study visit the next day. Participants are offered a paper version of the satiety questionnaire if they so desire. The satiety questionnaire asks the participants to evaluate their feelings of hunger, fullness, desire to eat, and satisfaction with the previous meal. Desire to eat is differentiated to the participant as a desire to consume food regardless of their state of hunger while satisfaction is differentiated from fullness to the participants as a psychological sensation of contentedness and not a physical sensation of fullness. The same questionnaire is used for all time points during each study visit. Participants are asked to refrain from consuming caffeine in the morning. A specific arrival time is set for arrival at the Innovation Center the following day between 8 and 8:40 AM.

After the subject arrives at the IU-Bloomington Innovation Center, coolers and icepacks are collected, compliance with the study protocol is confirmed. Next the diet record is reviewed by study personnel. Participants may be asked to clarify entries made on the diet record.

Participants are invited to a room where as many as 3 participants at a time will undergo the study protocol. Subjects are allowed to interact with each other but are instructed to refrain from discussing the snack bars. A baseline satiety questionnaire is completed before the snack bars are offered with a bottle of water. Participants are instructed to enter "1" with regard to satisfaction with the meal at this fasted time point. Ad libitum water intake is allowed throughout the study visit. The participants are instructed to consume two snack bars comprising 300 kcal as quickly and comfortably as possible. After the subjects consume the bars, study personnel provide the participant with a sensory evaluation, either printed or electronic, which asks the subject to evaluate the bars in terms of overall taste, sweetness, saltiness, savory, desire to eat more, with the meal, and fullness/satiation. Participants complete the sensory evaluation after having consumed both bars. If participants are unable to consume both bars, the sensory evaluation is not completed, and the experimental protocol is terminated for that subject.

The subjects remain in the room are are allowed bathroom breaks, to entertain themselves with their own audio devices, to read, and to work. Participants are prohibited from bringing and consuming outside food and from exercising during the study protocol. Satiety questionnaires are completed every 30 minutes from fasting. An electronic timer is provided with a flow sheet denoting the times for the satiety questionnaires to be completed. Participants write the times that they completed each iteration of the satiety questionnaire. Participants are monitored periodically for compliance and electronic recording of the questionnaires is monitored.

After 2 hours the penultimate satiety questionnaire for the study visit is completed. Subjects are informed that they will be escorted to a lunch buffet consisting of grilled hamburger patties, grilled chicken, brioche buns, sliced tomatoes, sliced medium cheddar cheese, mayonnaise, mustard and ketchup, a fruit tray with individual portions of watermelon, cantaloupe, strawberries and blueberries, a bowl of potato chips, a bowl of mixed, salted nuts, chocolate chip cookies, and whipped cream to add to any of the food they choose. Participants are instructed to "serve themselves as much of the food as they care to consume and to consume it until comfortably full as quickly and comfortably as possible." Participants log the time that they finished the meals and complete a final satiety questionnaire after lunch. Each food item is weighed by study personnel before and after the participants dine.

A second study visit is conducted that mirrors the first with a different type of snack bar. Start times for the protocol and the buffet lunch are matched as closely to the first study visit as possible.

ELIGIBILITY:
Inclusion Criteria:

* Persons 18 to 65 years of age, inclusive
* BMI 18.5-29.9 kg/m2 inclusive
* Subject understands the study procedures and signs forms documenting informed consent to participate in the study and is willing and able to complete study procedures.
* Subject is judged by the Co-Investigator to be in general good health without diabetes, cardiovascular disease, or cancer that has not been in remission in the past 3 years on the basis of medical history and screening measurements.
* Subject is willing and able to find their own transportation to the IU SPH metabolic kitchen for meal pickups and study visits.
* Subject can comply with study food consumption and energy intake during each treatment condition and access to safe storage and preparation of the provided dinner.
* Subject is willing to follow his/her usual physical activity throughout the study.

Exclusion Criteria:

* Subject is unwilling or unable to safely store, prepare (heat in a microwave oven), and consume the provided dinner meals and to control energy intake on the lead-in days.
* Subject is unable to comply with the study timeline.
* Because one of the dietary interventions contains eggs and whey, vegans and vegetarians who do not consume eggs or milk products are excluded. Lacto-ovo vegetarians are eligible to apply for participation.
* Subjects reporting allergies to any ingredients listed on the ingredient lists of each snack bar are not eligible. It should be noted that eggs, tree and ground nuts, and dairy appear on the ingredient lists and are examples (non-exhaustive) of common allergens that might disqualify a participant. The ingredient lists for each product is provided as an attachment.
* Subject is using medications known to affect appetite, blood lipids, body composition, body weight, or food intake such as statins and GLP-1 receptor agonists.
* Subject has a previous history of eating or gastrointestinal disorders such as Inflammatory Bowel Disease, Irritable Bowel Syndrome, Celiac Disease, gluten intolerance, stomach ulcers etc.
* Subject has had any form of bariatric surgery.
* Subject is currently known to be pregnant or is lactating.
* Subject has diagnosed metabolic diseases such as diabetes, cardiovascular disease such as hypertriglyceridemia, untreated hypercholesterolemia, or hypertension, that limits their intake of certain foods that may impact their health, or cancer within the last 3 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Food Intake | 2:15-2:30 minutes postprandial
  An individual buffet is provided in which participants consume as much food as they like until comfortably full. Buffet items include hamburgers, grilled chicken, buns, tomatoes, cheese, condiments (mayonnaise, mustard and ketchup), potato chips, mixed nuts, cookes, and a fruit tray of cantaloupe, watermelon, blueberries, strawberries, and pineapple with whipped cream offered as a condiment. Food are weighed before and after consumption of the buffet and macronutrient content is assessed from the nutrient facts label or from the USDA FoodData Central database.
Hunger | Fasting and every 30 minutes for 2 hours (5 time points)
  The study will assess hunger using 1-100 point visual analogue scales.
Fullness | Fasting and postprandial every 30 minutes for 2 hours (5 time points) at visits 1 and 2.
  The study will assess fullness using 1-100 point visual analogue scales.
Desire to eat | This question will be presented at fasting and postprandially every 30 minute for 2 hours (5 time points) at visit 1 and visit 2.
  The study will assess subjective desire to eat using a 1-100 point visual analogue scale.
Satisfaction with the meal | Presented at fasting, and every 30 minutes postprandially for 2 hours during visit 1 and 2
  Satisfaction with the meal will be assessed using a 1-100 point visual analogue scale.

OTHER OUTCOMES:
Taste | The sensory evaluation is completed after consumption of the snack bars on visit 1 and visit 2.
  The study will utilize a Likert scale using: dislike a great deal, dislike somewhat, Neither like nor dislike, like somewhat, like a great deal.
Sweetness | The sensory evaluation is completed after the subjects consume the snack bars on visits 1 and 2.
  A four point Likert scale using: too sweet, just sweet enough, not too sweet, and needs to be sweeter.
Saltiness | The sensory evaluation is completed after the subjects consume the bars on visits 1 and 2.
  A four point Likert scale uses: too salty, just right, could use a little more, and could use a lot more.
Bitterness | The sensory evaluation is completed following consumption of the snack bars on visits 1 and 2.
  A four point Likert scale is employed using: really bitter, not too bitter, very little bitterness, and no bitterness whatsoever.
Savoriness | Savoriness will be assessed after the subjects complete the snack bars on visits 1 and 2.
  A five point Likert scale will assess savoriness using: no savoriness whatsoever, very little savoriness, neither savory nor not savory, a little savory, and very savory.
Desire to consume more of this food | The sensory evaluation takes place after the subjects consume the snack bars at visit 1 and visit 2.
  A 1-100 point visual analogue scale will be used to assess the participants' desire to consume more of each product with the qualifiers "definitely not" at the low end and "definitely yes" on the high end of the visual analogue scale.
Fullness/satiation | The sensory evaluation takes place after the participants have consumed the snack bars on visits 1 and 2.
  Participants will assess their subjective feelings of fullness and satiation following consumption of the snack bars using a 1-100 point visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University--Bloomington School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
There is no need to share individual participant data.

REFERENCES:
- See also: This site provides a lay description of the study protocol and a link to a prescreening questionnaire for interested and potentially eligible individuals. — https://iu.co1.qualtrics.com/jfe/form/SV_6zKPV31WA6zO7z0